CLINICAL TRIAL: NCT04350541
Title: Heart Failure Associated With Chronic Obstructive Lung Disease and Maximum Exercise Tolerance: Evaluation of the Distribution and Pulmonary Deposition of Radioaerosol, Peripheral and Coronary Endothelial Function, Brain Natriuretic Peptide
Brief Title: Effects of HIIT in Tolerance to Exercise of Individuals With HF and Coexisting COPD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to COVID-19 pandemic
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, BRUNA THAYS SANTANA DE ARAÚJO, physiotherapist, clinical research, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07640919.4.0000.5208
Record Dates: First submitted 2020-03-23; First posted 2020-04-17 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval training (Experimental): Interval training will consist of 10 minutes of warm-up between 40-50% of the peak oxygen consumption (VO2peak), followed by four to six repetitions of three-minute intervals between 80-90% of VO2peak and three minutes between 40-50% VO2peak and finally, five minutes of cooling down between 30-40% of VO2peak.
  Interventions: Other: High-intensity interval training
- Continuous training (Active Comparator): The continuous aerobic training will consist of 10 minutes of warm-up with intensity between 40 and 50% of VO2peak, 20 minutes of conditioning between 60 and 70% of VO2peak and 5 minutes of cooling down between 30 and 40% of VO2peak.
  Interventions: Other: Continuous aerobic training

INTERVENTIONS:
Other: High-intensity interval training — Exercise with high-intensity intervals followed by active rest
  Arms: Interval training
Other: Continuous aerobic training — Interval Moderate-intensity aerobic training without intervals
  Arms: Continuous training

SUMMARY:
INTRODUCTION: The complexity of the pathophysiology of heterogeneous diseases such as heart failure and obstructive pulmonary disease causes a different approach to these diseases or with a view as much as a better understanding of the same situations, with which the clinical profile of patients who are associated with an association is. It is known that regular physical training promotes progressive improvements in exercise tolerance, in the pulmonary ventilation / perfusion ratio and in respiratory function by strengthening. OBJECTIVE: To compare the effects of high-intensity interval training and continuous aerobic exercise, with peripheral endothelial function, brain natriuretic peptide levels, maximum exercise tolerance, distribution of lung volumes and quality of life of patients with obstructive pulmonary disease associated with heart failure. METHODS: This is a clinical, controlled, randomized and blinded trial. Peripheral endothelial function, tolerance to maximum and submaximal exercise, distribution of lung volumes, quality of life, presence of symptoms of depression and perception of clinical change will be evaluated. EXPECTED RESULTS: Incorporate into the care of these patients, new effective therapeutic approaches, of low cost and with greater technical and scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals with Heart Failure of all etiologies;
* Diagnosed moderate and severe chronic obstructive pulmonary disease;
* Clinical stability;
* No change in the medication class within three months before the beginning of the research.

Exclusion Criteria:

* Unstable angina;
* Myocardial infarction;
* Previous cardiac surgery up to three months before the beginning of the study;
* Hemodynamic instability;
* Orthopedic and neurological diseases;
* Psychological and/or mental impairment.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | 24 weeks
  Evaluated by the cardiopulmonary exercise test by measuring the maximum oxygen consumption.
Peripheral endothelial function | 24 weeks
  Evaluated by the peripheral arterial tonometry using the EndoPat 2000 device

SECONDARY OUTCOMES:
Quality of life assessment: Short Form-36 questionnaire | 24 weeks
  Evaluated by the Short Form-36 questionnaire
Perception of clinical change | 24 weeks
  Evaluated by the Patient Global Impression of Change Scale which is a one-dimensional measure in which individuals can rate their associated improvement on a 7-item scale ranging from "1 = no changes" to "7 = much better".
Distance covered in the six-minute walk test | 24 weeks
  Evaluated by the six-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No